CLINICAL TRIAL: NCT02657473
Title: Long-term Inhaled Nebulized Tobramycin in Patients With Non-cystic Fibrosis Bronchiectasis. A Randomized Placebo Controlled Trial. The BATTLE Study Bronchiectasis And Tobramycin SoluTion InhaLation ThErapy.
Brief Title: Inhaled Nebulized Tobramycin in Non-cystic Fibrosis Bronchiectasis
Acronym: BATTLE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, W.G.Boersma, Dr.MD., Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54939
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Non-CF Bronchiectasis
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: . In present study the value of maintenance TIS will be investigated in patients with non-CF bronchiectasis colonized by different bacterial species sensitive for tobramycin.
  Objective: The primary outcome of the study is a 50% reduction in exacerbation rate in patients using maintenance TIS (OD). Secondary outcome parameters are lung function (FEV1, FVC), QoL (QOL-B), LTRI-VAS, Leicester cough score, bacterial load in sputum and tobramycin resistant pathogens.
  Study design: A randomised, double blind placebo controlled, multicenter study. Study population: Patients aged ≥ 18-year-old with confirmed bronchiectasis by (HR)CT and at least two exacerbations during previous 12 months.
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- TIS 300mg once daily (Active Comparator): Tobramycin inhalation solution (TIS) 300mg once daily for at least 9 months and up to 12 months
  Interventions: Drug: tobramycin inhalation solution
- Placebo once daily (Placebo Comparator): Saline 0.9% inhalation solution 300mg once daily for at least 9 months and up to 12 months
  Interventions: Drug: Saline 0.9% inhalation solution

INTERVENTIONS:
Drug: tobramycin inhalation solution
  Arms: TIS 300mg once daily
Drug: Saline 0.9% inhalation solution
  Arms: Placebo once daily

SUMMARY:
The purpose of this study is to evaluate the effect of tobramycin inhalation solution (TIS) once daily compared tot placebo in patients with non-CF bronchiectasis. The primary endpoint is a reduction of exacerbations of the disease during the treatment period. Next to this parameter the investigators expect to show a significant beneficial effect on lung function parameters, QoL, bacterial load of pathogens in sputum and tobramycin resistance.

DETAILED DESCRIPTION:
See uploaded study protocol

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. The presence of chronic respiratory symptoms such as cough, dyspnoea, expectoration of sputum
3. Confirmed non-CF bronchiectasis by (HR)CT
4. Documented history of at least 2 pulmonary exacerbations treated with courses of antibiotics within 12 months before inclusion.
5. No course of antibiotics or maintenance antibiotics (except for macrolides) 1 month prior to the start of the study.
6. Minimal one documented sputum or BAL-fluid culture with gram-negative bacteria or S.aureus within 12 months.
7. Growth of protocol defined pathogens in sputum at screening visit sensitive to tobramycin
8. Tolerance of inhaled tobramycin

Exclusion Criteria:

1. Any exacerbation within the month prior to the start of the study
2. Diagnosis of cystic fibrosis
3. Active allergic bronchopulmonary aspergillosis (ABPA)
4. Any oral, IV or inhaled antibiotics (except for macrolides) within 1 month prior to the start of the study
5. Any IV or IM corticosteroids or change in oral corticosteroids (> 10 mg) within 1 month prior to the start of the study
6. Any change/start treatment regimens macrolides, hypertonic saline, inhaled mannitol or other mucolytics, corticosteroids within 1 month prior to the start of the study
7. Change in physiotherapy technique or schedule within 1 month prior to the start of the study
8. Severe immunosuppression or active malignancy
9. Active tuberculosis
10. Chronic renal insufficiency (eGFR < 30 ml/min), use of loop diuretics
11. Have received an investigational drug or device within 1 month prior to the start of the study
12. Serious or active medical or psychiatric illness
13. Pregnancy and child bearing
14. History of poor cooperation or non-compliance
15. Unable to use nebulizers
16. Allergic for tobramycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-08-13 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Wim G. Boersma, Dr.MD, Principal Investigator — Medical Center Alkmaar
Locations (6):
- Netherlands (6):
  - North West Clinics, Alkmaar, North Holland
  - VU Medical Center, Amsterdam
  - Zuyderland Medisch Centrum, Heerlen
  - Spaarne Gasthuis, Hoofddorp
  - Canisius Ziekenhuis, Nijmegen
  - UMCU, Utrecht

REFERENCES:
- [Derived] Terpstra LC, Altenburg J, Bronsveld I, Doodeman HJ, Rozemeijer W, Heijerman HGM, Boersma WG. The BATTLE study: Effects of long-term tobramycin inhalation solution (TIS) once daily on exacerbation rate in patients with non-cystic fibrosis bronchiectasis. Study protocol of a double blind, randomized, placebo-controlled trial: study protocol. Contemp Clin Trials Commun. 2022 Dec 6;30:101045. doi: 10.1016/j.conctc.2022.101045. eCollection 2022 Dec. PMID 36531900
- [Derived] Terpstra LC, Altenburg J, Bronsveld I, de Kruif MD, Berk Y, Snijders D, Rozemeijer W, Heijerman HGM, Boersma WG. Effects of long-term tobramycin inhalation solution (TIS) once daily on exacerbation rate in patients with non-cystic fibrosis bronchiectasis. Respir Res. 2022 Dec 3;23(1):330. doi: 10.1186/s12931-022-02243-y. PMID 36463180

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02657473/Prot_SAP_000.pdf